CLINICAL TRIAL: NCT01722149
Title: Phase I Study for the Adoptive Transfer of Re-directed FAP-specific T Cells in the Pleural Effusion of Patients With Malignant Pleural Mesothelioma.
Brief Title: Re-directed T Cells for the Treatment (FAP)-Positive Malignant Pleural Mesothelioma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FAPME-1
Record Dates: First submitted 2012-10-31; First posted 2012-11-06 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: malignant pleural mesothelioma; re-directed T cells; FAP; fibroblast activation protein; CD8 positive T cells; pleural effusion
MeSH Terms: conditions — Mesothelioma, Malignant; Pleural Effusion

STUDY DESIGN:
Intervention Model Description: Adoptive Transfer of re-directed FAP-specific T cells
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adoptive Transfer of re-directed T cells (Experimental): Adoptive Transfer of re-directed FAP specific T cells in the pleural effusion
  Interventions: Genetic: Adoptive Transfer of re-directed T cells

INTERVENTIONS:
Genetic: Adoptive Transfer of re-directed T cells — Adoptive Transfer of 10e6 re-directed T cells in the pleural effusion

SUMMARY:
MPM patients are not eligible for surgical procedures like decortication or pleuro-pneumectomy and have a median survival of 12 months with palliative chemotherapy. Therefore, new therapeutic approaches are of crucial need in this clinical situation. This is a phase I trial for patients with malignant pleural mesothelioma with pleural effusion testing the safety of a fixed single dose of 1x10e6 adoptively transferred FAP-specific re-directed T cells given directly in the pleural effusion. Lymphocytes will be taken 21 days before transfer from peripheral blood. CD8 positive T cells will be isolated and re-programmed by retroviral transfer of a chimeric antigen receptor (CAR) recognizing FAP which serves as target structure in MPM.

* Trial with immunomodulatory product / biological

DETAILED DESCRIPTION:
This is a phase I trial for patients with malignant pleural mesothelioma. A fixed single dose of adoptively transferred FAP-specific CD8 positive re-directed T cells will be given in the pleural effusion.

Three patients who are at the time point of screening not operable will be treated with re-directed T cells administered into the pleural effusion after completion of 3 cycles of palliative chemotherapy. In the case of one AE grade III/IV or one SAE - and the occurrence of DLT both judged to be treatment related by an independent safety monitoring board - the patient number will be expanded to 6 patients. The study will be stopped if one additional DLT occurs also judged to be treatment related.

Patients will be treated with 1x10e6 re-directed FAP-specific T cells injected in the pleural effusion. The study ends 35 days after adoptive T cell transfer. Re-directed FAP-specific T cells will be administered at day 0 (day 14 of the third cycle of palliative chemotherapy). The study is designed to demonstrate safety of 1x10e6 re-directed FAP-specific T cells. The next patient will be enrolled earliest, when the previous patient completed day +14 and the safety monitoring board has not declared any DLTs. The palliative chemotherapy is not part of the study protocol.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed and documented malignant pleural mesothelioma with pleural effusion,
* Signed Informed Consent after being informed,
* Patients medically and/or functionally at screening not accessible for surgical treatment
* Bone marrow function: hemoglobin >/= 100 g/L; white blood cell count (WBC) >/= 1.0 x 109/L; absolute neutrophile count (ANC) >/= 0.5 x 109/L; platelet count >/= 100 x 109/L,
* Hepatic: aspartate transaminase (AST) and alanine transaminase (ALT) </= 2.5 times upper limit of normal (ULN)); bilirubin </= 1.5 x ULN,
* Renal: creatinine = 176 umol/l and creatinine clearance = 45 mL/min,
* No concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents,
* The patient has received no major organ allograft,
* HIV-negative,
* HBV and HCV negative,
* No uncontrolled bleeding disorder,
* Patients of child-producing potential must agree to use contraception while enrolled in the study and for 24 months after the adoptive transfer.

Exclusion criteria:

* Contra-indications to the class of TpP, e.g. known hypersensitivity or allergy to the investigational product,
* Contra-indications on ethical grounds,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception: Safe contraception is defined as follows:Female and male subjects of childbearing potential, using and willing to continue using a medically reliable method of double barrier contraception for the entire study duration and the next 2 years, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices in combination with preservatives. Or subjects who are using any other method considered sufficiently reliable by the investigator in individual cases.Subjects who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Known or suspected non-compliance, drug or alcohol abuse
* Pericardial effusion of more than 100 ml. Pericardial involvement assessed by CT scan
* Patients with medical history of coronary heart disease (CHD), stroke or peripheral vascular disease (PVD),
* Patients with medical history of autoimmune disease such as multiple sclerosis, lupus, rheumatoid arthritis, inflammatory bowel disease or small vessel vasculitis,
* Regular intake of immune-modulating drugs,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Safety | until 35 days after transfer of re-directed T cells
  Incidence and severity of treatment-related laboratory abnormalities, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version v4.03 criteria as grade III-IV. In the case of one AE grade III/IV or one SAE the safety monitoring board will judge whether the case is treatment related and whether it have to be counted as DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Curioni, MD, Principal Investigator — University Hospital Zurich, Division of Oncology
Locations (1):
- University Hospital Zurich, Division of Oncology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Schuberth PC, Hagedorn C, Jensen SM, Gulati P, van den Broek M, Mischo A, Soltermann A, Jungel A, Marroquin Belaunzaran O, Stahel R, Renner C, Petrausch U. Treatment of malignant pleural mesothelioma by fibroblast activation protein-specific re-directed T cells. J Transl Med. 2013 Aug 12;11:187. doi: 10.1186/1479-5876-11-187. PMID 23937772
- [Background] Petrausch U, Schuberth PC, Hagedorn C, Soltermann A, Tomaszek S, Stahel R, Weder W, Renner C. Re-directed T cells for the treatment of fibroblast activation protein (FAP)-positive malignant pleural mesothelioma (FAPME-1). BMC Cancer. 2012 Dec 22;12:615. doi: 10.1186/1471-2407-12-615. PMID 23259649